CLINICAL TRIAL: NCT03504436
Title: Evaluation of the LEO + Stent in the Endovascular Treatment of Wide Neck Intracranial Aneurysms (Fusiform, Saccular or Dissecting), Ruptured or Not Ruptured: Cohort of the Self-expanding Intracranial Stent LEO
Brief Title: Endovascular Treatment of Wide Neck Intracranial Aneurysms With the LEO + Stent : The LEO + II Cohort Study
Status: Completed | Type: Observational
Sponsor: Balt Extrusion (Industry)
Responsible Party: Sponsor
Other Study IDs: LEO + II
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2018-04

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: LEO + — LEO +: self-expanding intracranial stent

SUMMARY:
This is a prospective, multicenter, single-arm observational study to evaluate the efficacy and the morbi-mortality of LEO + in patients with wide neck intracranial aneurysms (fusiform, saccular or dissecting), ruptured or not ruptured.

ELIGIBILITY:
Inclusion Criteria:

* All patients with ruptured or not ruptured intracranial aneurysms demonstrated by cerebral arteriography treated with LEO + stent
* Patients (or their parents for minors) must be informed and give written consent

Exclusion Criteria:

* Patients (or parents) who refused to give consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with ruptured or not ruptured intracranial aneurysms demonstrated by cerebral arteriography treated with LEO + stent
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2015-03-15 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Total aneurysmal occlusion rate | 18 months
  Classification of the occlusion observed angiographically as "complete occlusion", "residual neck" or "residual aneurysm" using the Montreal three-grade scale
Morbi-mortality | 18 months
  Number of complications and/or device or procedure related adverse events

IPD SHARING:
Plan to Share IPD: No